CLINICAL TRIAL: NCT00092339
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose Study to Evaluate the Effects of Rofecoxib 50 mg and Valdecoxib 40 mg in Patients With Postoperative Dental Pain
Brief Title: A Study of Two Approved Drugs in the Treatment of Postoperative Dental Pain (0966-190)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0966-190; 2004_069
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Pain
Keywords: dental surgery; molar removal
MeSH Terms: conditions — Pain, Postoperative | interventions — rofecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0966, rofecoxib
Drug: Comparator: valdecoxib, placebo

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of two approved drugs in the treatment of pain following dental surgery.

DETAILED DESCRIPTION:
The duration of treatment is 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Impaction of a molar tooth requiring removal

Exclusion Criteria:

* Any known allergy to the study drugs

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2002-08-01 (Actual); Primary Completion 2002-09-15 (Actual); Study Completion 2002-09-15 (Actual)

PRIMARY OUTCOMES:
Overall analgesic effect as measured by total pain relief over 12 hours.

SECONDARY OUTCOMES:
Overall analgesic effect over 8 hrs.
Time to onset of analgesic, peak analgesic and duration of analgesic effects.
Percent of patients using and amount used of supplemental analgesia within 8, 12, and 24 hrs.
Overall safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Daniels SE, Desjardins PJ, Bird SR, Smugar SS, Tershakovec AM. Rofecoxib 50 mg and valdecoxib 20 or 40 mg in adults and adolescents with postoperative pain after third molar extraction: results of two randomized, double-blind, placebo-controlled, single-dose studies. Clin Ther. 2006 Jul;28(7):1022-34. doi: 10.1016/j.clinthera.2006.07.005. PMID 16990080
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html